CLINICAL TRIAL: NCT04171128
Title: Procalcitonin Role in Influenza Patients With Regard to Morbidity, Mortality and Antibiotic Use
Status: Completed | Type: Observational
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: AB3420-3
Record Dates: First submitted 2019-11-14; First posted 2019-11-20 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Influenza
Keywords: procalcitonin
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: antibiotic stewardship efforts — The local antibiotic team plan to implement procalcitonin use among the hospital physicians. the interventions are not ready yet.

SUMMARY:
The investigators intend to observe the inflammatory marker procalcitonin (PCT) in comparison with patient variables on morbidity, mortality and antibiotic treatment.

The overall aim is to observe if a low PCT value can have potential in reducing unessesary antibiotic use in seasonal influenza patients.

DETAILED DESCRIPTION:
This is an observational study of the clinical utility of early PCT measurements in seasonal influenza, with particular attention to PCT's predictive value for prognosis and bacterial respiratory superinfection. The aim is to evaluate PCT as a supplementary aid in the standard clinical evaluation of influenza patients. Patients may be included if a positive influenza test is reported within 48 hours after an initial clinical suspicion of influenza, and the hospital stay is lasting more than one day. The investigators have included 74 patients from the second half of the 2018-19 influenza season and will continue to include patients from the complete 2019-20 season.

Primary endpoints: Mortality (in-hospital and within 30 days post-discharge), bacterial respiratory tract superinfection.

Secondary endpoints: Intensive care unit stay, the proportion of patients on antibiotic use and total antibiotic use in doses and LOT ("length-of-treatment").

ELIGIBILITY:
Inclusion Criteria:

* patient admitted to the hospital with positive influenza test

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: seasonal influenza patients, adult population
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
mortality | 30 days
  From the national registry the investigators will register wheather or not the patient has died within day 14 and day 30, and in case of dead the date will be registered

SECONDARY OUTCOMES:
antibiotic use | up to one year
  From a elecronical medical chart (Metavision) the investigators will search and register the type of antibiotic used, the days of treatment and the total dose given in grams

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid christensen, MD, Principal Investigator — Ostfold hospital trust, Kalnes
Locations (2):
- Norway (2):
  - Ostfold Hospital trust, Sarpsborg, Akershus
  - Ostfold Hospital Trust, Sarpsborg, Østfold fylke

IPD SHARING:
Plan to Share IPD: No